CLINICAL TRIAL: NCT01164358
Title: Long Term Observation of Patient Satisfaction Post INTRACOR Treatment Based on Patient Perception and Diagnostic Data
Status: Completed | Type: Observational
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 1002
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Presbyopia
Keywords: Presbyopia; INTRACOR; patient satisfaction; long term
MeSH Terms: conditions — Presbyopia; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- study arm I: patients who have been enrolled in the previous study "Intrastromal Correction of Ametropia by Femtosecond Laser (study ISCAF), study arm 1, Presbyopia sub-group: treatment pattern 5-Rings"
- study arm II: patients who have been enrolled in the previous study "Intrastromal Presbyopia Correction by Means of Femtosecond Laser (study # 0905)"

SUMMARY:
This study is a prospective, open, not randomized, unilateral multicenter eye study consisting of two study arms to observe the long term satisfaction of patients after an INTRACOR treatment. The satisfaction is determined with the help of the patient perception and the subjective / objective diagnostic data.

The hypothesis of the study is that patients after an INTRACOR treatment are satisfied in the long term.

DETAILED DESCRIPTION:
The study is divided into two study arms. The first study arm includes patients of the preceding study "Intrastromal Correction of Ametropia by Femtosecond Laser (study ISCAF), study arm 1, Presbyopia sub-group: treatment pattern 5-Rings" and the second study arm includes patients of the previous "Intrastromal Presbyopia Correction by Means of Femtosecond Laser (study # 0905)".

The hypothesis of the study is that patients after a INTRACOR treatment are satisfied in the long term.

By detailed patient information and a clarification conversation it is guaranteed that every interested and agreeing patient fulfils the inclusion criteria of this study. The quantitative measuring values of the patient perception are assessed by a questionnaire. For measuring the subjective / objective diagnostic data only certificated diagnostic devices are used. No invasive intervention in the eye will be made to change the visual acuity.

Within the scope of the study between 98 and 135 patients should be examined. 49 to 63 patient are intended for the first study arm and 49 to 72 for the second study arm.

The follow-up examinations are carried out at 12 months and/or 24 months as well as for 36 months after the INTRACOR treatment. The study end points are determined for all follow-up examinations. The aim criteria should be reached for the final examination, which is after 36 months, at the latest.

ELIGIBILITY:
Inclusion Criteria:

* Age: at least 18 years old
* Patients must have read, understood and signed the Patient Information
* Patients are willing and able to return for follow-up examinations
* Patient has been already enrolled in the previous study "Intrastromal Correction of Ametropia by Femtosecond Laser (study ISCAF), study arm 1, Presbyopia sub-group: treatment pattern 5-Rings" or "Intrastromal Presbyopia Correction by Means of Femtosecond Laser (study # 0905)"

Exclusion Criteria:

* Continual wearing of contact lenses before the follow-up examination . Patients must refrain from wearing contact lenses for at least 14 days prior to these dates
* Patients who are pregnant or are lactating
* Patients who are participating in another ophthalmological clinical study except "Intrastromal Presbyopia Correction by Means of Femtosecond Laser (study # 0905)"
* severe sick people who cannot give any information on their visual acuity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Just patients who have been already enrolled in the previous study "Intrastromal Correction of Ametropia by Femtosecond Laser (study ISCAF), study arm 1, Presbyopia sub-group: treatment pattern 5-Rings" or "Intrastromal Presbyopia Correction by Means of Femtosecond Laser (study # 0905)"
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
long term satisfaction of patients post INTRACOR treatment based on a questionnaire | 36 months
  Satisfaction is assesed by three questions:
  Do you fell comfortable with the treatment result? Would you do the traetment again? Would you recommend the treatment to a relativ or a friend?
  If two out of these three questions are answered with "yes" then it can be assumed that the patient is satisfied.

SECONDARY OUTCOMES:
Determination if there is any correlation between patient satisfaction and subjective/objective diagnostic data. | 36 months
  Objective: Change in topographic map Subjective: uncorrected near visual acuity, uncorrected distance visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Mike P. Holzer, Prof. Dr. med, Principal Investigator — University of Heidelberg, department Ophthalmology
Locations (4):
- Germany (4):
  - University of Heidelberg, department Ophthamology, Heidelberg, Baden-Wurttemberg
  - FreeVis LASIK Center Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - Augenklinik am Marienplatz AG & Co. KG, Munich, Bavaria
  - ye-clinic for Refractive and Ophthalmo-Surgery, EJK Niederrhein, Duisburg, North Rhine-Westphalia

REFERENCES:
- [Derived] Thomas BC, Fitting A, Khoramnia R, Rabsilber TM, Auffarth GU, Holzer MP. Long-term outcomes of intrastromal femtosecond laser presbyopia correction: 3-year results. Br J Ophthalmol. 2016 Nov;100(11):1536-1541. doi: 10.1136/bjophthalmol-2015-307672. Epub 2016 Feb 22. PMID 26903524